CLINICAL TRIAL: NCT02894892
Title: Intragastric pH and Bismuth Effect for H. Pylori Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 201512127MINC
Record Dates: First submitted 2016-07-27; First posted 2016-09-09 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2016-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Electron Microscopy; Helicobacter pylori; Bismuth
MeSH Terms: interventions — bismuth phosphate, copolymers of vinyl acetate, dichlorophen, propionyl-acetophenone, triethanolamine, vinyl chloride, vinylisobutyl ether, zinc oxide drug combination; boron-doped bismuth oxybromide; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- (A)Bismuth (Active Comparator): (A)Bismuth (120mg/tab) 1 dose prior 1 hr before endoscopy
  Interventions: Drug: (A)Bismuth
- (B)Bismuth (Active Comparator): (B)Bismuth (120mg/tab) 1 dose in the morning and endoscopy in the afternoon
  Interventions: Drug: (B)Bismuth
- (C)Bismuth (Active Comparator): (C)Bismuth (120mg/tab) q.i.d. and endoscopy the next day
  Interventions: Drug: (C)Bismuth
- (D)Esomeprazole and Bismuth (Active Comparator): (D)3 days esomeprazole (40mg/tab) q.i.d. followed by bismuth (120mg/tab) 1 dose prior 1 hr before endoscopy
  Interventions: Drug: (D)Esomeprazole and Bismuth
- (E)Esomeprazole and Bismuth (Active Comparator): (E)3 days esomeprazole (40mg/tab) q.i.d. followed by bismuth (120mg/tab) 1 dose in the morning and endoscopy in the afternoon
  Interventions: Drug: (E)Esomeprazole and Bismuth
- (F)Esomeprazole and Bismuth (Active Comparator): (F)3 days esomeprazole (40mg/tab) q.i.d. followed by bismuth (120mg/tab) q.i.d. and endoscopy the next day
  Interventions: Drug: (F)Esomeprazole and Bismuth
- (G)Control (Other): (G)These patients underwent endoscopy due to abdominal discomfort or other symptoms and did not have cancers in the digestive tract after series of workup.
  Interventions: Other: (G)Control

INTERVENTIONS:
Drug: (A)Bismuth
  Other Names: (A)Active Comparator-Bismuth
  Arms: (A)Bismuth
Drug: (B)Bismuth
  Other Names: (B)Active Comparator-Bismuth
  Arms: (B)Bismuth
Drug: (C)Bismuth
  Other Names: (C)Active Comparator-Bismuth
  Arms: (C)Bismuth
Drug: (D)Esomeprazole and Bismuth
  Other Names: (D)Active Comparator-Esomeprazole and Bismuth
  Arms: (D)Esomeprazole and Bismuth
Drug: (E)Esomeprazole and Bismuth
  Other Names: (E)Active Comparator-Esomeprazole and Bismuth
  Arms: (E)Esomeprazole and Bismuth
Drug: (F)Esomeprazole and Bismuth
  Other Names: (F)Active Comparator-Esomeprazole and Bismuth
  Arms: (F)Esomeprazole and Bismuth
Other: (G)Control
  Other Names: (G)Other-Control
  Arms: (G)Control

SUMMARY:
Gastric cancer is one of the leading causes of cancer-related deaths worldwide. In Taiwan, there are around 3800 fresh cases annually, with about 5% of total cancers cases. Gastric cancer development is known to follow a multistate process from non-atrophic gastritis, atrophic gastritis, intestinal metaplasia, dysplasia, and carcinoma; H. pylori infection plays the key role of this carcinogenic process. Although H. pylori eradication would result in a marked gastric cancer reduction, treatment success using standard regimens has become more difficult in recent years, and increased antibiotic resistance is considered the most important reason for decreased treatment efficacy. As no specific new medications have been introduced in recent years, novel treatment regimens have been created using different combinations, durations and sequences of available medications. The addition of bismuth improved the cure rates despite a high prevalence of resistance, and resistance of H. pylori to bismuth has not been reported. Bismuth absorption is not required for efficacy in H. pylori treatment regimens, suggesting a local mechanism of action. The mechanisms of bismuth with responsible for rapid destruction of H. pylori within the stomach remain unclear. Knowledge of the mechanism of action of bismuth compounds against H. pylori would be beneficial in the development of improved treatment regimens in this era of declining eradication success rates. We conduct the pilot study to evaluate the bacteria fragments of H. pylori in specimen through electron microscopy after bismuth therapy and provide insight into the mechanism of action of pH on bismuth therapy. We also help to develop optimal H. pylori therapeutic strategies.

ELIGIBILITY:
Inclusion criteria

1. Age 20-69
2. Confirmed H. pylori infection by urea breath test or previous histology
3. Scheduled endoscopy
4. Mentally competent to be able to understand the consent form for individuals equal to or older than 20
5. Able to communicate with study staff for individuals equal to or older than 20
6. Without history of gastric cancer Exclusion criteria

1.History of gastric cancer

Deferral criteria:

1. Having received antibiotic treatment in the previous 15 days
2. Need of time to decide participation

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
The morphological changes of post-drug H. pylori by electron microscopy. | 3 years
  Endoscopy: The biopsy procedure protocol specified sampling gastric mucosa in the locations of gastric antrum, body and cardia (two specimens from each location). Specimens would be sent for electron microscopy.
  Electron microscopy: Bacteria fragments of H. pylori would be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsien Chiang, MD, M.Sc., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan